CLINICAL TRIAL: NCT05212233
Title: Financial Difficulty in Patients With Blood Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Boston University (Other); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 2063
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MM and/or CLL: This is a non-interventional study. All enrolled patients will complete a telephone interview. A subset of patients will complete the optional follow-up interview. The clinical practice sites through which patients are being recruited and enrolled on to the study will each complete the Site Survey. Physicians at these sites who treat patients with MM or CLL will be invited to complete the Physician Survey.

SUMMARY:
This is a hypothesis-driven, observational, cross-sectional, multi-site study of the financial difficulties experienced by patients undergoing treatment for multiple myeloma (MM) and chronic lymphocytic leukemia (CLL). It is composed of a patient survey (n=250) (Appendix A), a physician survey (n=100) (Appendix B), and a practice survey completed by each site enrolling patients onto this study (Appendix C). A subset of enrolled patients (n=35) will be invited to participate in an optional second telephone interview (Appendix D). This study will measure the prevalence of patient-reported financial difficulty, specific financial burdens and resources currently available to patients and from practices to assist with patient financial navigation.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVES:

To estimate the proportion of individuals with MM and/or CLL who report experiencing financial difficulty in the past 12 months.

SECONDARY OBJECTIVES:

Our seventeen secondary objectives address ten aspects of patient financial experience of cancer treatment:

Financial difficulty

2.2.1 To describe the association of patient report of financial difficulty with patient reported racial identity.

2.2.2 To describe the association of patient report of financial difficulty with insurance status.

Financial navigation

2.2.3 To describe the association of patient report of financial difficulty with receiving treatment at practices that report offering patients financial guidance through navigators or social workers, and with socioeconomic status.

2.2.4 To describe the current resources dedicated to patient financial navigation at participating sites, and types of psychosocial, transportation and financial navigation interventions sites are developing.

Financial burden

2.2.5 To identify distinct patterns of financial burden among patients undergoing treatment for MM and/ or CLL.

2.2.6 To examine the relationship between distinct patterns of financial burden with patient report of financial difficulty, and with patient sociodemographic, disease and treatment characteristics.

Financial support

2.2.7 To estimate the proportion of patients with MM and/or CLL undergoing treatment who report receiving financial support in the past 12 months.

2.2.8 To describe the association of patient report of receiving financial support with receiving treatment at practices offering patients financial guidance through navigators or social workers, and with socioeconomic status.

Patient concerns regarding treatment and costs of care

2.2.9 To describe the magnitude of patient concerns regarding treatment and costs of care.

2.2.10 To describe the association of patient concerns regarding treatment and costs of care with patient sociodemographic, disease and treatment characteristics, and practice characteristics.

Patient health and well-being

2.2.11 To describe the association of financial difficulty with patient self-reported health and well-being.

Physician discussion of financial difficulties with patients

2.2.12 To estimate the proportion of individuals with MM and CLL who have received treatment in the past 12 months and report to their physician experiencing financial difficulties related to their cancer care.

2.2.13 To identify the types of financial difficulties related to cancer care that patients discuss with their provider and care team.

Physician attitudes regarding patient communication about financial difficulties

2.2.14 To describe physician attitudes or preferences for how they or the care team discuss financial difficulties with patients.

Physician use of resources for addressing financial difficulties

2.2.15 To describe the resources used by physicians and their care team to help address patient reported financial difficulties related to cancer care.

Physician perspective on the impact of COVID-19 on patient financial difficulties

2.2.16 To assess COVID-19 related disruptions to physicians' practice with respect to addressing financial difficulties in patients.

Patient experience of financial difficulties

2.2.17 To conduct semi-structured qualitative interviews with a subset of patients to elucidate the patient experience of financial difficulties over time and its impact on cancer care, and structural barriers to accessing care and/or financial assistance.

ELIGIBILITY:
Inclusion Criteria:

PATIENT ELIGIBILITY CRITERIA

* Patients must have current diagnosis of chronic lymphocytic leukemia (CLL) or multiple myeloma (MM)
* Patients' medical records must be available to the registering institution
* Eligible patients must have been prescribed drug-based anticancer therapy, whether administered orally or by infusion, within the prior 12 months. Specifically, eligible patients are those who:

  * Are presently being treated with infused or orally-administered anticancer therapy, OR
  * Completed infused or orally-administered anti-cancer therapy in the past 12 months, OR
  * Were prescribed infused or orally-administered anticancer therapy within the prior 12 months yet chose to forego treatment
* Not currently enrolled in a clinical trial in which drug is supplied by the study
* Patients with psychiatric illness or other mental impairment that would preclude their ability to give informed consent or to respond to the telephone survey are not eligible
* Patients must be able to read and comprehend English or Spanish

SITE ELIGIBILITY CRITERIA

* Intent to complete the Practice Survey
* Access to patient medical records: Registering institution must have access to patient medical records, either on site or via request from other institutions, if recruiting patients at a site (as medical abstraction is required for collecting study data).
* Sites seeking to enroll Spanish- speaking patients must have Spanish speaking staff on site or through the use of a translation service to be able to conduct the informed consent discussion in Spanish.

PHYSICIAN ELIGIBILITY CRTERIA

* The physician currently treats patients with chronic lymphocytic leukemia (CLL) and/or multiple myeloma (MM).
* The physician is a treating physician at a site which has opened this protocol (LCCC 2063) and/or a site which opened the Alliance protocol (A231602CD; ClinicalTrials.gov Identifier: NCT03870633). Eligible physicians do not need to have their own patients enrolled onto this protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a current diagnosis of CLL or MM, prescribed drug-based anticancer therapy in the prior 12 months, with medical records available to the registering institution and who speak English or Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of patients with MM and/or CLL who report experiencing financial difficulty in the past 12 months. | Cross-sectional study / Baseline
  Financial difficulties will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) financial difficulty item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?", measured as "Not at all/A little/Quite a bit/Very much." Participant responses will be dichotomized as follows: "Not at all" or "A little" classified as "No", and "Quite a bit" and "very much" classified as "Yes." This dichotomized response will be assessed using Wilson score confidence interval (95%).

SECONDARY OUTCOMES:
To describe the association of patient report of financial difficulty with patient reported racial identity. | Cross-sectional study / Baseline
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) financial difficulty item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?", measured as "Not at all/A little/Quite a bit/Very much." Participant responses will be dichotomized as follows: "Not at all" or "A little" classified as "No", and "Quite a bit" and "very much" classified as "Yes." Will be assessed using Mann-Whitney U test and logistic regression.
To describe the association of patient report of financial difficulty with insurance status. | Cross-sectional study / Baseline
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) financial difficulty item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?", measured as "Not at all/A little/Quite a bit/Very much." Participant responses will be dichotomized as follows: "Not at all" or "A little" classified as "No", and "Quite a bit" and "very much" classified as "Yes." Will be assessed using Mann-Whitney U test and logistic regression.
To describe the association of patient report of financial difficulty with receiving treatment at practices that report offering patients financial guidance through navigators or social workers, and with socioeconomic status. | Cross-sectional study / Baseline
  Assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) financial difficulty item #28 regarding financial difficulties with a modified recall period: "Has your physical condition or medical treatment caused you financial difficulties in the past year?", measured as "Not at all/A little/Quite a bit/Very much." Participant responses will be dichotomized as follows: "Not at all" or "A little" classified as "No", and "Quite a bit" and "very much" classified as "Yes." Will be assessed logistic regression and latent class analysis models with covariates.
To describe the current resources dedicated to patient financial navigation at participating sites, and types of psychosocial, transportation and financial navigation interventions sites are developing. | Cross-sectional study / Baseline
  Assessed using site-reported plans of current resources and developing psychosocial, transportation and financial navigation services found in a Practice Survey
To identify distinct patterns of financial burden among patients undergoing treatment for MM and/or CLL. | Cross-sectional study / Baseline
  Assessed using patient reported difficulties paying medical bills (4 binary items), delays or foregoing treatment (4 binary items), difficulties covering non-medical expenses due to costs of treatment (2 binary items), and financial worries (5 binary items)
To examine the relationship between distinct patterns of financial burden with patient report of financial difficulty, and with patient sociodemographic, disease and treatment characteristics. | Cross-sectional study / Baseline
  Assessed using patient reported difficulties paying medical bills (4 binary items), delays or foregoing treatment (4 binary items), difficulties covering non-medical expenses due to costs of treatment (2 binary items), and financial worries (5 binary items)
To estimate the proportion of patients with MM and/or CLL undergoing treatment who report receiving financial support in the past 12 months. | Cross-sectional study / Baseline
  The proportion of patients who report receiving financial support (patient survey part 2 question 3 [yes/no]) in the past 12 months will be described using summary statistics.
To describe the association of patient report of receiving financial support with receiving treatment at practices offering patients financial guidance through navigators or social workers, and with socioeconomic status. | Cross-sectional study / Baseline
  Logistic regression with receipt of financial support in the past 12 months (patient survey part 2 question 3 [yes/no]) as the dependent variable will be used to test the hypothesis that individuals with multiple myeloma (MM) or chronic lymphocytic leukemia (CLL) will be more likely to report receipt of financial support if they are treated at practices reporting that they offer patients financial guidance through navigators or social workers compared to those treated at practices without these resources. The model will control for disease/treatment characteristics and indicators of patient socioeconomic status.
To describe the magnitude of patient concerns regarding treatment and costs of care. | Cross-sectional study / Baseline
  Aggregate scores of the Valuing Dimensions of the Patient Experience Questionnaire measuring patient concerns regarding treatment and costs of care (part 1, questions 22-36 of the protocol patient survey) will be analyzed descriptively. These questions are all assessed as "Very worried", "Somewhat worried" and "Not worried" will be scored as 2, 1 and 0 respectively and aggregated using standard practices.
To describe the association of patient concerns regarding treatment and costs of care with patient sociodemographic, disease and treatment characteristics, and practice characteristics. | Cross-sectional study / Baseline
  Aggregate scores of the Valuing Dimensions of the Patient Experience Questionnaire measuring patient concerns regarding treatment and costs of care (part 1, questions 22-36 of the protocol patient survey) will be stratified by demographics (e.g. gender, race/ethnicity), socioeconomic characteristics (e.g. education, income), disease characteristics (e.g. MM, CLL), and practice-specific factors (e.g. presence of a social worker/patient navigator). These questions are all assessed as "Very worried", "Somewhat worried" and "Not worried" will be scored as 2, 1 and 0 respectively and aggregated using standard practices. Differences in the aggregate scores between groups will be tested using t-tests. Adjustment for multiple comparisons will not be conducted, which is consistent with social science and/or preference based research.
To describe the association of financial difficulty with patients self-reported health and well-being. | Cross-sectional study / Baseline
  Aggregate scores of the PROMIS-10 and EQ-5D-5L will be utilized as covariates in a logistic regression model to assess if there is any association with them and the outcome of patient-reported financial difficulty (item #28 of the EORTC QLQ-C30). The PROMIS-10 is a 10-item instrument scored on a scale from 0 - 50 (higher scores = improved QOL). The EQ-5D-5L is a 5-item instrument (5 point scales scored 1-5, where higher scores = worse QOL) and the EQ Visual Analogue scale to score the patient's self-rated health on a scale from 0-100, where higher scores = better QOL.
To estimate the proportion of individuals with MM and CLL who have received treatment in the past 12 months and report to their physician experiencing financial difficulties related to their cancer care. | Cross-sectional study / Baseline
  Assessed through a physician survey (Likert scale percentage categories) described using summary statistics.
To identify the types of financial difficulties related to cancer care that patients discuss with their provider and care team. | Cross-sectional study / Baseline
  Assessed through a physician survey (Likert scale percentage categories) described using summary statistics.
To describe physician attitudes or preferences for how they or the care team discuss financial difficulties with patients. | Cross-sectional study / Baseline
  Assessed through a physician survey (Likert scale percentage categories) described using summary statistics.
To describe the resources used by physicians and their care team to help address patient reported financial difficulties related to cancer care. | Cross-sectional study / Baseline
  Resources provided to patients (Likert scale responses), and changes in these resources in past 12 months (questions 13-15) (Open text and ordered categorical) assessed via a physician survey. Described using summary statistics of ordered categorical responses and qualitative summary of open text responses
To assess COVID-19 related disruptions to physicians' practice with respect to addressing financial difficulties in patients. | Cross-sectional study / Baseline
  Physician Survey, 2 questions (multiple choice and open text and ordered categorical responses). Described using summary statistics of ordered categorical responses and qualitative summary of open text responses
To conduct semi-structured qualitative interviews with a subset of patients to elucidate the patient experience of financial difficulties over time and its impact on cancer care, and structural barriers to accessing care and/or financial assistance. | Cross-sectional study / Within 8 weeks after Patient Survey is completed
  Assessed using a semi-structured qualitative interview guide. Interview transcripts will be coded thematically. Emergent themes will be summarized and illustrated with exemplar quotes.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Bennett, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (7):
- United States (7):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Albert Einstein College of Medicine, The Bronx, New York
  - UNC Medical Center, Chapel Hill, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials